CLINICAL TRIAL: NCT00986180
Title: A Randomized, Double-Blind, Parallel-Group Study of NUCYNTA (Tapentadol) Immediate Release vs. Oxycodone Immediate Release for the Treatment of Acute Low Back Pain
Brief Title: NUCYNTA (Tapentadol Immediate Release) Versus Oxycodone Immediate Release in the Treatment of Acute Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR015643; R331333PAI3025 (Other: Ortho-McNeil Janssen Scientific Affairs, LLC); KF5503/51 (Other: Grünenthal)
Record Dates: First submitted 2009-09-25; First posted 2009-09-29 (Estimated); Results first posted 2012-02-29 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Pain; Back Pain; Low Back Pain; Back Pain With Radiation
Keywords: Acute Low Back Pain; Low Back Pain With Leg Pain Below The Knee; Radiculopathy, Oxycodone; Tapentadol; NUCYNTA
MeSH Terms: conditions — Pain; Back Pain; Low Back Pain; Radiculopathy | interventions — Tapentadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Experimental): NUCYNTA 50 75 or 100 mg every 4 to 6 hours for up to 10 days as needed for pain
  Interventions: Drug: NUCYNTA
- 002 (Active Comparator): Oxycodone IR 5 10 or 15 mg every 4 to 6 hours for up to 10 days as needed for pain
  Interventions: Drug: Oxycodone IR

INTERVENTIONS:
Drug: NUCYNTA — 50, 75, or 100 mg every 4 to 6 hours for up to 10 days as needed for pain
  Arms: 001
Drug: Oxycodone IR — 5, 10, or 15 mg every 4 to 6 hours for up to 10 days as needed for pain
  Arms: 002

SUMMARY:
Evaluate how NUCYNTA (tapentadol) immediate release (IR) compares with oxycodone IR in the treatment of acute low back pain.

DETAILED DESCRIPTION:
This is a randomized, outpatient, multicenter, double-blind study (blinded to patient and to study doctor) comparing NUCYNTA to oxycodone IR in the treatment of patients with acute (new onset) low back pain who also have associated leg pain that radiates (travels down) below the knee. Patients will be screened for study eligibility at Visit 1. The study will be explained and informed consent will be obtained. Potential patients must satisfy all eligibility criteria to be enrolled in the study. Eligible candidates will proceed to the Double-Blind Treatment Phase. At the time of study entry, all prohibited medications will be discontinued and will be disallowed throughout the study. All patients will call into an interactive voice response system (IVRS) to complete a pain assessments twice daily throughout the study. Patients who discontinue early for any reason will be instructed to contact the study site to complete final assessments, prior to taking supplemental pain medication if applicable, and to schedule a final study visit. All patients will return to the study site on Day 5 (Visit 2) where they will be evaluated by study personnel and, as appropriate, continue with study treatment for an additional 5 days. Patients will return to the study site for the final visit on Day 10/End of Study (Visit 3) when they will have all final study assessments. The treatment duration will be up to 10 days. The sponsor will collect adverse events starting with the signing of the informed consent form. Adverse events will be reported by the subject for the duration of the study. Any clinically significant abnormalities persisting at the end of the study will be followed by the investigator until resolution or until a clinically stable endpoint is reached. Blood samples for serum chemistry and hematology and a urine sample for urinalysis will be collected. The investigator will review the laboratory report, document this review, and record any clinically relevant changes occurring during the study. The following tests will be performed by the central laboratory: Urine Pregnancy Testing for women of childbearing potential only, Urine Drug Screen, Vital Signs (pulse rate and blood pressure), Physical Examination, Neurological Examination, and Vomiting Assessment. The study will be conducted at approximately 80 sites in the United States (US). Patients will be randomized to one of the two following treatment groups: NUCYNTA 50, 75 or 100 mg every 4 to 6 hours up to 10 days as needed for pain. Oxycodone IR 5, 10 or 15 mg every 4 to 6 hours as needed for pain. Patients will begin treatment on Day 1 with one "lower dose" capsule of study drug (NUCYNTA 50 mg or oxycodone IR 5 mg). Subsequent dose adjustments will be made by study patients, as needed, to achieve a dose that provides a meaningful improvement in their pain intensity

ELIGIBILITY:
Inclusion Criteria:

* At Visit 1 (study entry) patients must have a medical history and physical and neurological examinations that support a clinical diagnosis of acute low back pain that is felt down to the lower leg below the knee with the onset no longer than 30 days before Visit 1
* At Visit 1 patients must report qualifying pain intensity scores
* Patients must be appropriate candidates for treatment with oral opioid pain medication in the investigator's clinical judgment
* Patients must be able to appropriately verbalize pain characteristics and to complete all protocol required measurements/assessments without assistance
* Patients must be medically stable on the basis of physical examination, medical history, vital signs, and clinical laboratory tests performed at screening

Exclusion Criteria:

* History of back (cervical, thoracic or lumbosacral) pain =50% of the time in the 1 year prior to the first visit
* History of any low back pain episode, with the exception of the current acute low back pain episode, within 3 months prior to the first visit that was greater than mild in pain intensity, or was associated with disability (e.g., loss of time from work, family, or activities of daily living), or necessitated the use of an opioid (narcotic) analgesic including tramadol
* Medical history or physical examination results that suggest the acute low back pain or any of the neurological symptoms or signs are caused by a serious medical condition (e.g., fever, chills, unexplained weight loss, bowel or urinary bladder dysfunction or incontinence, bilateral leg weakness, progressive weakness, paralysis)
* There is a high probability for surgical intervention for the back pain during the projected time on the study or that there will be an increase in the severity of the leg pain or deficits
* Had either a surgical procedure involving the spine or intervertebral discs in the lower back region within 1 year prior to Visit 1 or had >1 surgical procedure(s) involving the spine or intervertebral discs in the lower back region
* has any painful condition that could interfere with the study assessments or with the patient's ability to differentiate the pain associated with the acute low back pain episode from pain associated with another condition
* History of severe lumbar spinal stenosis, fibromyalgia, or ankylosing spondylitis
* history of epilepsy or recurrent seizures
* Unable or unwilling to discontinue all prohibited medications at the time of randomization and during the time of their participation in the study
* Known or suspected history of alcohol or drug abuse based on medical history, physical examination, urine drug screening, or the investigator's clinical judgment
* History of cancer malignancy within 2 years prior to the first visit, with the exception of basal cell skin carcinoma
* Have filed or plan to file a worker's compensation claim for any issue related to the current acute low back pain episode
* Currently involved in litigation or plan to seek legal recourse for any issue related to their acute low back pain
* Known allergies, hypersensitivity, or intolerance to tapentadol or the comparator (oxycodone) or any excipients used in their manufacture
* Had previously been enrolled in a tapentadol clinical study
* is pregnant or are breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ortho-McNeil Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Ortho-McNeil Janssen Scientific Affairs, LLC
Locations (74):
- United States (74):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Jonesboro, Arkansas
  - Fresno, California
  - Garden Grove, California
  - Glendale, California
  - Laguna Hills, California
  - Palm Springs, California
  - Pismo Beach, California
  - Wildomar, California
  - Denver, Colorado
  - Fairfield, Connecticut
  - Boynton Beach, Florida
  - Clearwater, Florida
  - Edgewater, Florida
  - Jacksonville, Florida
  - Lake Worth, Florida
  - Miami, Florida
  - Newport Richey, Florida
  - Oldsmar, Florida
  - Pembroke Pines, Florida
  - Saint Cloud, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Savannah, Georgia
  - Avon, Indiana
  - Evansville, Indiana
  - Overland Park, Kansas
  - Lexington, Kentucky
  - Covington, Louisiana
  - Mandeville, Louisiana
  - Metairie, Louisiana
  - New Orleans, Louisiana
  - Sunset, Louisiana
  - Fall River, Massachusetts
  - North Dartmouth, Massachusetts
  - Kalamazoo, Michigan
  - Florissant, Missouri
  - Springfield, Missouri
  - Washington, Missouri
  - Henderson, Nevada
  - Pahrump, Nevada
  - Atco, New Jersey
  - Blackwood, New Jersey
  - Cherry Hill, New Jersey
  - North Massapequa, New York
  - Williamsville, New York
  - Charlotte, North Carolina
  - Hickory, North Carolina
  - Mooresville, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Andover, Ohio
  - Beavercreek, Ohio
  - Centerville, Ohio
  - Cincinnati, Ohio
  - Marion, Ohio
  - Oklahoma City, Oklahoma
  - Altoona, Pennsylvania
  - Tyrone, Pennsylvania
  - Murrells Inlet, South Carolina
  - Nashville, Tennessee
  - Austin, Texas
  - Bryan, Texas
  - Bulverde, Texas
  - Houston, Texas
  - Lake Jackson, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Clinton, Utah
  - Orem, Utah
  - Danville, Virginia

REFERENCES:
- [Derived] Biondi D, Xiang J, Benson C, Etropolski M, Moskovitz B, Rauschkolb C. Tapentadol immediate release versus oxycodone immediate release for treatment of acute low back pain. Pain Physician. 2013 May-Jun;16(3):E237-46. PMID 23703422

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 19 subjects either did not take medication or did not have verifiable drug exposure. 2 subjects were randomized in two different sites, information was included for only one site. 1 subject was randomized in error.
Groups:
- NUCYNTA: 50, 75 or 100 mg every 4 to 6 hours as needed for pain for up to 10 days; max daily dose 600 mg
- Oxycodone IR: 5, 10 or 15 mg every 4 to 6 hours as needed for pain for up to 10 days; max daily dose 90 mg
Period: Overall Study
Arm/Group | NUCYNTA | Oxycodone IR
Started | 321 | 324
Completed | 277 | 268
Not Completed | 44 | 56
Not completed — Adverse Event | 21 | 23
Not completed — Lack of Efficacy | 4 | 3
Not completed — Lost to Follow-up | 5 | 7
Not completed — Physician Decision | 1 | 3
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 1 | 9
Not completed — Miscellanies | 10 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NUCYNTA | Oxycodone IR | Total
Number analyzed (Participants) | 321 | 324 | 645
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 282 | 297 | 579
  >=65 years | 39 | 26 | 65
Age Continuous [Mean (Standard Deviation); unit: years] | 45.7 (14.18) | 45.1 (14.36) | 45.4 (14.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 176 | 321
  Male | 176 | 148 | 324
Region of Enrollment [Number; unit: participants]
  UNITED STATES | 321 | 324 | 645
Baseline Low Back Pain Intensity [Mean (Standard Deviation); unit: Units on a scale] — Pain intensity scale is: 0=no pain, 10=Pain as bad as you can imagine.
  Units on a scale | 7.2 (1.66) | 7.2 (1.54) | 7.2 (1.60)
Baseline Index Leg Pain Intensity [Mean (Standard Deviation); unit: Units on a scale] — Pain intensity scale is: 0=no pain, 10=Pain as bad as you can imagine.
  Units on a scale | 6.2 (2.21) | 6.2 (2.10) | 6.2 (2.15)
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 43 | 39 | 82
  Not Hispanic or Latino | 278 | 283 | 561
  Not Reported | 0 | 2 | 2
Baseline BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.9 (8.83) | 30.4 (8.63) | 30.6 (8.72)

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Difference (SPID) for Low Back Pain - Summary Statistics at 120 Hours (With Imputation)
Description: Pain intensity is an 11-point numerical rating scale (NRS). 0=no pain, 10=Pain as bad as you can imagine. The pain intensity difference (PID) was to be calculated as baseline pain minus current pain at each assessment time point. SPID is a weighted sum of PID over a specified time period, say 120 hours.
Time Frame: 0 hour (prior to first dose) and 120 hours
Population: Modified Intent-To-Treat Population: All randomized subjects who take at least 1 dose of study drug and have a baseline assessment of pain, and the baseline low back pain intensity assessment score ≥5 on an 11-point NRS (recorded via the IVRS).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 287 | 298
Units on a scale | 264.6 (11.43) | 264.0 (11.22)
Statistical Analysis 1: Comparison: NUCYNTA; Test type: Non-Inferiority or Equivalence — The sample size was recalculated due to Amendment INT-1. The non-inferiority margin for SPID120 was set as 120. The common standard deviation for the SPID120 data was estimated to be 230. Seventy nine subjects in each arm would have 90% power to demonstrate the non-inferiority of NUCYNTA to oxycodone IR with a 1-sided significance level of 0.025. This would have required enrollment of total 158 mITT subjects for each stratum. The original sample size (292 mITT subjects) was derived for SPID72; p = 0.9703, ANCOVA; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-32.1 to 30.9], Standard Error of Mean 16.02

2. Secondary Outcome: Sum of Pain Intensity Difference (SPID) for Low Back Pain - Summary Statistics at 2 Days (With Imputation)
Description: Pain intensity is an 11-point numerical rating scale (NRS). 0=no pain, 10=Pain as bad as you can imagine. The pain intensity difference (PID) was to be calculated as baseline pain minus current pain at each assessment time point. SPID is a weighted sum of PID over a specified time period, say 2 days.
Time Frame: Day 0 and Day 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 287 | 298
Units on a Scale | 80.1 (4.34) | 81.8 (4.26)
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; p = 0.7691, ANCOVA; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [-10.1 to 13.7], Standard Error of Mean 6.08

3. Secondary Outcome: SPID for Low Back Pain - Summary Statistics at 3 Days (With Imputation)
Description: Pain intensity is an 11-point numerical rating scale (NRS). 0=no pain, 10=Pain as bad as you can imagine. The pain intensity difference (PID) was to be calculated as baseline pain minus current pain at each assessment time point. SPID is a weighted sum of PID over a specified time period, say 3 days.
Time Frame: Day 0 and Day 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 287 | 298
Units on a scale | 137.2 (6.60) | 138.1 (6.47)
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; p = 0.9282, ANCOVA; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-17.3 to 19.0], Standard Error of Mean 9.24

4. Secondary Outcome: SPID for Low Back Pain - Summary Statistics at 10 Days (With Imputation)
Description: Pain intensity is an 11-point numerical rating scale (NRS). 0=no pain, 10=Pain as bad as you can imagine. The pain intensity difference (PID) was to be calculated as baseline pain minus current pain at each assessment time point. SPID is a weighted sum of PID over a specified time period, say 10 days.
Time Frame: Day 0 and Day 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 287 | 298
Units on a scale | 540.2 (21.23) | 538.6 (20.84)
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; p = 0.9562, ANCOVA; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-60.1 to 56.8], Standard Error of Mean 29.75

5. Secondary Outcome: SPID for Index Leg Pain - Summary Statistics at 2 Days (With Imputation)
Description: as for outcome 2
Time Frame: Day 0 and Day 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 287 | 298
Units on a Scale | 73.6 (4.34) | 72.1 (4.26)
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; p = 0.7973, ANCOVA; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-13.5 to 10.4], Standard Error of Mean 6.08

6. Secondary Outcome: SPID for Index Leg Pain - Summary Statistics at 3 Days (With Imputation)
Description: as for outcome 3
Time Frame: Day 0 and Day 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 287 | 298
Units on a Scale | 125.5 (6.63) | 123.0 (6.51)
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; p = 0.7882, ANCOVA; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-20.8 to 15.8], Standard Error of Mean 9.30

7. Secondary Outcome: SPID for Index Leg Pain - Summary Statistics at 5 Days (With Imputation)
Description: Pain intensity is an 11-point numerical rating scale (NRS). 0=no pain, 10=Pain as bad as you can imagine. The pain intensity difference (PID) was to be calculated as baseline pain minus current pain at each assessment time point. SPID is a weighted sum of PID over a specified time period, say 5 days.
Time Frame: Day 0 and Day 5
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 287 | 298
Units on a Scale | 239.2 (11.29) | 234.1 (11.08)
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; p = 0.7491, ANCOVA; Mean Difference (Final Values) = -5.1, 95% CI 2-sided [-36.1 to 26.0], Standard Error of Mean 15.82

8. Secondary Outcome: SPID for Index Leg Pain - Summary Statistics at 10 Days (With Imputation)
Description: as for outcome 4
Time Frame: Day 0 and Day 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 287 | 298
Units on a Scale | 488.0 (20.71) | 476.4 (20.33)
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; p = 0.6897, ANCOVA; Mean Difference (Final Values) = -11.6, 95% CI 2-sided [-68.6 to 45.4], Standard Error of Mean 29.03

9. Secondary Outcome: Total Pain Relief (TOTPAR) for Low Back Pain - Summary Statistics at 5 Days
Description: Pain Relief - 5-Point Numerical Rating Scale, 0=None, 4=Complete. Total Pain Relief (TOTPAR) is a weighted sum of pain relieve over a specified time period, say 5 days.
Time Frame: Day 0 and Day 5
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 287 | 298
Units on a Scale | 254.8 (5.01) | 256.4 (4.91)
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; p = 0.8226, ANCOVA; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-12.2 to 15.4], Standard Error of Mean 7.02

10. Secondary Outcome: SF-MPQ-2 - Change From Baseline Values: Subscale and Total Scores - Continuous Pain Day 5
Description: Short-Form McGill Pain Questionnaire - 2 (SF-MPQ-2) is a 22-question instrument. Each item lists different qualities of pain or related symptoms and is scored using an 11-point NRS ranging from (pain or symptom is not present) to 10 (worst possible pain). Subscale scores are calculated as the mean of the items in that subscale ranged from 0 to 10. Continuous pain subscale descriptors include: throbbing pain, cramping pain, gnawing pain, aching pain, heavy pain, and tender.
Time Frame: Day 0 and Day 5
Population: Intent-To-Treat Population (all randomized subjects who take at least 1 dose of study drug and have a baseline assessment of pain) and have both baseline and Day 5 SF-MPQ-2 measurement
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 274 | 276
Units on a Scale | -2.4 (2.05) | -2.4 (2.14)
Statistical Analysis 1: Comparison: NUCYNTA; Test type: Superiority or Other; p = 0.8880, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: SF-MPQ-2 - Change From Baseline Values: Subscale and Total Scores - Continuous Pain Day 10/Last Visit
Description: as for outcome 10
Time Frame: Day 0 and Day 10
Population: Intent-To-Treat Population and have both baseline and Day 10 SF-MPQ-2 measurements.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 289 | 298
Units on a Scale | -3.1 (2.35) | -2.9 (2.31)
Statistical Analysis 1: Comparison: NUCYNTA; Test type: Superiority or Other; p = 0.4115, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: SF-MPQ-2 - Change From Baseline Values: Subscale and Total Scores - Intermittent Pain Day 5
Description: Short-Form McGill Pain Questionnaire - 2 (SF-MPQ-2) is a 22-question instrument. Each item lists different qualities of pain or related symptoms and is scored using an 11-point NRS ranging from (pain or symptom is not present) to 10 (worst possible pain). Subscale scores are calculated as the mean of the items in that subscale ranged from 0 to 10. Intermittent pain subscale descriptors include: shooting pain, stabbing pain, sharp pain, splitting pain, electric-shock pain, and piercing.
Time Frame: Day 0 and Day 5
Population: Intent-To-Treat Population and have both baseline and Day 5 SF-MPQ-2 measurements.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 274 | 276
Units on a Scale | -2.6 (2.23) | -2.5 (2.09)
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; p = 0.8495, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: SF-MPQ-2 - Change From Baseline Values: Subscale and Total Scores - Intermittent Pain Day 10/Last Visit
Description: as for outcome 12
Time Frame: Day 0 and Day 10
Population: Intent-To-Treat Population and have both baseline and Day 10 SF-MPQ-2 measurements.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 289 | 298
Units on a Scale | -3.3 (2.46) | -3.2 (2.29)
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; p = 0.7846, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: SF-MPQ-2 - Change From Baseline Values: Subscale and Total Scores - Neuropathic Pain Day 5
Description: Short-Form McGill Pain Questionnaire - 2 (SF-MPQ-2) is a 22-question instrument. Each item lists different qualities of pain or related symptoms and is scored using an 11-point NRS ranging from (pain or symptom is not present) to 10 (worst possible pain). Subscale scores are calculated as the mean of the items in that subscale ranged from 0 to 10. Predominantly neuropathic pain subscale descriptors include: hot-burning pain, cold-freezing pain, pain caused by light touch, itching, tingling or "pins and needles" and numbness.
Time Frame: Day 0 and Day 5
Population: Intent-To-Treat Population and have both baseline and Day 5 SF-MPQ-2 measurements.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 274 | 276
Units on a Scale | -1.5 (1.92) | -1.4 (1.85)
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; p = 0.4790, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: SF-MPQ-2 - Change From Baseline Values: Subscale and Total Scores - Neuropathic Pain Day 10/Last Visit
Description: as for outcome 14
Time Frame: Day 0 and Day 10
Population: Intent-To-Treat Population and have both baseline and Day 10 SF-MPQ-2 measurements.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 289 | 298
Units on a Scale | -1.8 (1.94) | -1.6 (1.99)
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; p = 0.3147, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: SF-MPQ-2 - Change From Baseline Values: Subscale and Total Scores - Affective Descriptors Day 5
Description: Short-Form McGill Pain Questionnaire - 2 (SF-MPQ-2) is a 22-question instrument. Each item lists different qualities of pain or related symptoms and is scored using an 11-point NRS ranging from (pain or symptom is not present) to 10 (worst possible pain). Subscale scores are calculated as the mean of the items in that subscale ranged from 0 to 10. Affective subscale descriptors include: tiring-exhausting, sickening, fearful, and punishing-cruel.
Time Frame: Day 0 and Day 5
Population: Intent-To-Treat Population and have both baseline and Day 5 SF-MPQ-2 measurements.
Measure: Mean (Standard Deviation); unit: score of scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 274 | 276
score of scale | -2.0 (2.46) | -1.9 (2.31)
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; p = 0.5411, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: SF-MPQ-2 - Change From Baseline Values: Subscale and Total Scores - Affective Descriptors Day 10/Last Visit
Description: as for outcome 16
Time Frame: Day 0 and Day 10
Population: Intent-To-Treat Population and have both baseline and Day 10 SF-MPQ-2 measurements.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 289 | 298
Units on a Scale | -2.4 (2.74) | -2.2 (2.39)
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; p = 0.6137, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: SF-MPQ-2 - Change From Baseline Values: Subscale and Total Scores - Total Score Day 5
Description: Short-Form McGill Pain Questionnaire - 2 (SF-MPQ-2) is a 22-question instrument. Each item lists different qualities of pain or related symptoms and is scored using an 11-point NRS ranging from (pain or symptom is not present) to 10 (worst possible pain). The total SF-MPQ-2 scale score is calculated as the mean of all 22 items. The range of the total score is 0 to 10.
Time Frame: Day 0 and Day 5
Population: Intent-To-Treat Population and have both baseline and Day 5 SF-MPQ-2 measurements.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 275 | 277
Units on a Scale | -2.2 (1.84) | -2.1 (1.74)
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; p = 0.7246, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: SF-MPQ-2 - Change From Baseline Values: Subscale and Total Scores - Total Score Day 10/Last Visit
Description: as for outcome 18
Time Frame: Day 0 and Day 10
Population: Intent-To-Treat Population with both baseline and Day 10 SF-MPQ-2 measurements.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 290 | 298
Units on a Scale | -2.7 (2.04) | -2.5 (1.91)
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; p = 0.4882, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Patient Global Impression of Change at End of Study
Description: Patient Global Impression of Change (PGIC) assesses the subject's global improvement since starting study treatment using a 7-point NRS (1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse).
Time Frame: Day 0 and Day 10/last visit
Population: Intent-To-Treat Population.
Measure: Number; unit: Units on a Scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 302 | 311
Units on a Scale
  1 = Very much improved | 89 | 90
  2 = Much improved | 111 | 116
  3 = Minimally improved | 59 | 67
  4 = No change | 27 | 24
  5 = Minimally worse | 2 | 0
  6 = Much worse | 1 | 0
  7 = Very much worse | 1 | 1
  Missing | 12 | 13
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; p = 0.7201, Cochran-Mantel-Haenszel

21. Secondary Outcome: Patient Global Impression of Change at End of Study
Description: as for outcome 20
Time Frame: Day 0 and Day 10/lst visit
Population: Intent-To-Treat Population with PGIC assessment.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 290 | 298
Units on a Scale | 2.1 (1.04) | 2.1 (0.96)

22. Secondary Outcome: Clinician Global Impression of Change at End of Study
Description: Clinician Global Impression of Change (CGIC) assesses the subject's global improvement since starting study treatment using a 7-point NRS (1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse).
Time Frame: Day 0 and Day 10/last visit
Population: Intent-To-Treat Population.
Measure: Number; unit: Units on a Scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 302 | 311
Units on a Scale
  1 = Very much improved | 78 | 77
  2 = Much improved | 127 | 130
  3 = Minimally improved | 60 | 70
  4 = No change | 21 | 18
  5 = Minimally worse | 2 | 1
  6 = Much worse | 1 | 0
  7 = Very much worse | 2 | 0
  Missing | 12 | 13
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; p = 0.5208, Cochran-Mantel-Haenszel

23. Secondary Outcome: Clinician Global Impression of Change at End of Study
Description: as for outcome 22
Time Frame: Day 0 and Day 10/last visit
Population: Intent-To-Treat Population with CGIC assessment.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 290 | 298
Units on a Scale | 2.1 (0.99) | 2.1 (0.93)

24. Secondary Outcome: Satisfaction With Treatment at Day 5
Description: The subject's satisfaction with treatment was assessed using a 7-point scale (1=Very satisfied, 2=Somewhat satisfied, 3=Slightly satisfied, 4=Neither satisfied nor dissatisfied, 5=Slightly dissatisfied, 6=Somewhat dissatisfied, 7=Very dissatisfied).
Time Frame: Day 0 and Day 5
Population: Intent-To-Treat Population.
Measure: Number; unit: Units on a Scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 302 | 311
Units on a Scale
  1 = Very satisfied | 113 | 92
  2 = Somewhat satisfied | 102 | 132
  3 = Slightly satisfied | 31 | 32
  4 = Neither satisfied nor dissatisfied | 16 | 5
  5 = Slightly dissatisfied | 8 | 7
  6 = Somewhat dissatisfied | 2 | 5
  7 = Very dissatisfied | 3 | 4
  Missing | 27 | 34
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; p = 0.0401, Cochran-Mantel-Haenszel

25. Secondary Outcome: Satisfaction With Treatment at Day 5
Description: as for outcome 24
Time Frame: Day 0 and Day 5
Population: Intent-To-Treat Population with subject's satisfaction assessment on Day 5.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 275 | 277
Units on a Scale | 2.0 (1.19) | 2.0 (1.18)

26. Secondary Outcome: Satisfaction With Treatment at End of Study
Description: as for outcome 24
Time Frame: Day 0 and Day 10/last visit
Population: Intent-To-Treat Population.
Measure: Number; unit: Units on a Scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 302 | 311
Units on a Scale
  1 = Very satisfied | 146 | 148
  2 = Somewhat satisfied | 84 | 87
  3 = Slightly satisfied | 28 | 29
  4 = Neither satisfied nor dissatisfied | 7 | 14
  5 = Slightly dissatisfied | 7 | 3
  6 = Somewhat dissatisfied | 8 | 4
  7 = Very dissatisfied | 10 | 13
  Missing | 12 | 13
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; p = 0.4679, Cochran-Mantel-Haenszel

27. Secondary Outcome: Satisfaction With Treatment at End of Study
Description: as for outcome 24
Time Frame: Day 0 and Day 10/last visit
Population: Intent-To-Treat Population with subject's satisfaction assessment at end of the study.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 290 | 298
Units on a Scale | 2.0 (1.49) | 2.0 (1.48)

28. Secondary Outcome: Incidence of 30% Responders Without Nausea or Vomiting at Day 5
Description: Number of subjects had ≥ 30% reduction from baseline in low back pain intensity without nausea or vomiting reported.
Time Frame: Day 0 and Day 5
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 287 | 298
Participants | 117 | 104
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; p = 0.1454, Fisher Exact

29. Secondary Outcome: Incidence of 50% Responders Without Nausea or Vomiting at Day 5
Description: Number of subjects had ≥ 50% reduction from baseline in low back pain intensity without nausea or vomiting reported.
Time Frame: Day 0 and Day 5
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 287 | 298
Participants | 72 | 60
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; p = 0.1541, Fisher Exact

30. Secondary Outcome: Summary of Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation
Time Frame: Day 0 and Day 10/last visit
Population: Safety Population: all randomized subjects who take at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 321 | 324
Participants
  Number of subjects with adverse events | 21 | 26
  Eye disorders | 1 | 0
  Vision blurred | 1 | 0
  Gastrointestinal disorders | 11 | 14
  Nausea | 6 | 9
  Vomiting | 5 | 6
  Diarrhea | 1 | 1
  Abdominal discomfort | 1 | 0
  Constipation | 0 | 1
  General disorders and admin. site conditions | 2 | 0
  Fatigue | 2 | 0
  Infections and infestations | 0 | 1
  Upper respiratory tract infection | 0 | 1
  Injury, poisoning and procedural complications | 0 | 1
  Contusion | 0 | 1
  Investigations | 1 | 1
  Hepatic enzyme increased | 1 | 0
  Liver function test abnormal | 0 | 1
  Musculoskeletal and connective tissue disorders | 2 | 1
  Back pain | 1 | 1
  Muscle spasms | 1 | 0
  Neoplasms benign, malignant and unspecified | 1 | 0
  Lung cancer metastatic | 1 | 0
  Nervous system disorders | 6 | 9
  Dizziness | 3 | 3
  Somnolence | 2 | 2
  Headache | 1 | 2
  Convulsion | 0 | 1
  Syncope | 0 | 1
  Psychiatric disorders | 0 | 1
  Depression | 0 | 1
  Skin and subcutaneous tissue disorders | 1 | 3
  Rash | 0 | 2
  Pruritus | 0 | 1
  Rash generalized | 1 | 0

31. Secondary Outcome: Summary of Subjects Having Nausea as a Treatment-Emergent Adverse Event
Description: Number of subjects that reported nausea as a treatment-emergent adverse event during the study.
Time Frame: Day 0 and Day 10/last visit
Population: Safety Population: all randomized subjects who take at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 321 | 324
Participants | 51 | 67
Statistical Analysis 1: Comparison: NUCYNTA; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.92 to 2.06]

32. Secondary Outcome: Summary of Subjects Having Vomiting as a Treatment-Emergent Adverse Event
Description: Number of subjects that reported vomiting as a treatment emergent adverse event during the study.
Time Frame: Day 0 and Day 10/last visit
Population: Safety Population: all randomized subjects who take at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 321 | 324
Participants | 51 | 80
Statistical Analysis 1: Comparison: NUCYNTA; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.74, 95% CI 2-sided [1.17 to 2.57]

33. Secondary Outcome: Summary of Subjects Having Constipation as a Treatment-Emergent Adverse Event
Description: Number of subjects that reported constipation as a treatment emergent adverse event during the study.
Time Frame: Day 0 and Day 10/last visit
Population: Safety Population: all randomized subjects who take at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 321 | 324
Participants | 7 | 23
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.43, 95% CI 2-sided [1.45 to 8.11]

34. Secondary Outcome: Summary of Subjects Having Pruritus as a Treatment-Emergent Adverse Event
Description: Number of subjects that reported pruritus as a treatment emergent adverse event during the study.
Time Frame: Day 0 and Day 10/last visit
Population: Safety Population: all randomized subjects who take at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 321 | 324
Participants | 27 | 26
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.54 to 1.67]

35. Secondary Outcome: Kaplan-Meier First Time to 30% Response From Baseline for Low Back Pain
Description: 30% response means >= 30% reduction from baseline in low back pain intensity score.
Time Frame: Day 0 and Day 10/last visit
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 287 | 298
Hours | 42.93 [33.83 to 48.97] | 44.27 [30.72 to 54.97]
Statistical Analysis 1: Comparison: NUCYNTA vs Oxycodone IR; Test type: Superiority or Other; p = 0.5828, Log Rank

36. Secondary Outcome: Kaplan-Meier First Time to 50% Response From Baseline for Low Back Pain
Description: 50% response means >= 50% reduction from baseline in low back pain intensity score.
Time Frame: Day 0 and Day 10/last visit
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | NUCYNTA | Oxycodone IR
Number analyzed (Participants) | 287 | 298
Hours | 92.05 [71.93 to 107.92] | 107.45 [78.65 to 127.38]
Statistical Analysis 1: Comparison: NUCYNTA; Test type: Superiority or Other; p = 0.9084, Log Rank

ADVERSE EVENTS:
Arm/Group | NUCYNTA | Oxycodone IR
Serious Adverse Events (participants affected / at risk) | 2/321 | 3/324
Other Adverse Events (participants affected / at risk) | 141/321 | 165/324
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NUCYNTA (N=321) | Oxycodone IR (N=324)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NUCYNTA (N=321) | Oxycodone IR (N=324)
Nausea (Gastrointestinal disorders) | 51 | 67
Vomiting (Gastrointestinal disorders) | 51 | 80
Constipation (Gastrointestinal disorders) | 7 | 23
Dizziness (Nervous system disorders) | 38 | 34
Somnolence (Nervous system disorders) | 26 | 22
Headache (Nervous system disorders) | 14 | 20
Pruritus (Skin and subcutaneous tissue disorders) | 27 | 26

LIMITATIONS AND CAVEATS:
There were 19 subjects either did not take medication or did not have verifiable drug exposure. 2 subjects were randomized in two different sites, only one site information were included. 1 subject were randomized in error.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days